CLINICAL TRIAL: NCT05207930
Title: GAmified HOme-based COgnitive-Nutritional Training (GAHOCON) for Older People With Cognitive Frailty: A Feasibility Study
Brief Title: GAmified HOme-based COgnitive-Nutritional Training Feasibility Study
Acronym: GAHOCON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah College (Other); Mindvivid (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-UAMH
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Frailty; Protective Diet Adherence; Cognitive Function; Frailty; Nutrition; Body Composition
Keywords: Cognitive frailty; Randomized controlled trial; Nutrition; Protective diets; Gamification; Home-based intervention
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: A total of 40 eligible subjects will be randomly assigned into 2 groups, with block sizes of 8 people in a ratio of 1:1. The intervention group will undertake a 4-week centre-based training followed by an 8-week home-based gamified cognitive-nutrition training (i.e., GAHOCON). Meanwhile, the control group will also receive the same 4-week centre-based training. Afterwards, the control group will be introduced to some open-source cognitive game and will be encouraged to participate in these games in the elderly centre. In other words, the control will not receive the GAHOCON treatment at all.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors at both pre- and post-observations will be blinded to the group label.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This arm will undertake a centre-based health education on nutrition and cognitive frailty for 4 weeks, followed by an 8-week homed based gamified cognitive-nutrition training (GAHOCON).
  Interventions: Device: GAmified HOme-based COgnitive-Nutrition training (GAHOCON)
- Control Group (Placebo Comparator): This arm will undertake the same centre-based health education on nutrition and cognitive frailty for 4 weeks but will be opened to undertake a remotely supervised online open-source cognitive games, with which the contents are unrelated to nutrition, at the elderly community centre.
  Interventions: Device: Centre-based online open-source cognitive games

INTERVENTIONS:
Device: GAmified HOme-based COgnitive-Nutrition training (GAHOCON) — A home-based tablet game training, in which participants are expected to apply the nutrition knowledge they learn from the centre-based nutritional education and their cognitive functions.
  Participants in the intervention group are expected to engage in the home-based training regularly during those 8 weeks. A team of registered social workers working in the elderly community centre will monitor the progress, remind, set goals, and provide supports to the participant remotely on WhatsApp.
  Arms: Intervention Group
Device: Centre-based online open-source cognitive games — During the 8 weeks in which the intervention group receives GAHOCON treatment, the control group will be introduced to some online open-source cognitive games (e.g. CogniFit) and are encouraged to play those games at the elderly community centre. However, the content of these games are unrelated to nutrition and the training is gamified to a less extent compared to GAHOCON. They will have free access to these online open-source cognitive games at the elderly community centre.
  Arms: Control Group

SUMMARY:
Background: Cognitive frailty is an at-risk state of dementia that it can be reversed by manipulating the lifestyle factors, such as cognitive activity and nutrition/dietary pattern. Their protective effects depend on a prolonged adherence to these factors. However, in the literature, most of the cognitive interventions are centred-based and supervised. Nutrition intervention depends on the provision of supplement or a complimentary supply of food. There is a lack of interventions with components of sustaining cognitive and nutrition training effect for the community-dwelling older people with cognitive frailty in home settings.

Objectives: This study aims to examine the feasibility and preliminary effects of a gamified, home-based, cognitive-nutritional training (GAHOCON) programme for community-dwelling older people with cognitive frailty on protective diet adherence, cognitive function, frailty nutrition, and body composition.

DETAILED DESCRIPTION:
Methods: This study employs a pilot randomized controlled trial design. Recruitment will be conducted in elderly community centres. Participants who are aged ≥ 60 years, community-dwelling, and having cognitive frailty will be recruited. Participants will be randomized into either intervention or control group at a 1:1 ratio by permuted block randomization with a block size of 8 people. In the intervention group, participants will attend both centre-based training for one month and home-based training for 2 months. Health education on cognitive frailty and nutrition are included in the centre-based training. GAHOCON is included in the home-based training. The gamified cognitive-nutritional training employs digital gaming technology to develop a programme by combining cognitive training and nutrition education to promote the health of older people cognitive frailty. In the control group, participants will attend only the centre-based training. For the outcomes, this study will measure the feasibility in terms of the willingness of participants to be randomized, study participation rate, follow-up rates, response rates to questionnaires, adherence rate, level of participation of the tablet-based training, and time needed for data collection. Adherence to protective diets, cognitive function, frailty, nutrition, and body composition will be measured at baseline (T0), immediately after the completion of the intervention (T1). Convenience sampling will be employed to recruit 30-40 subjects for pilot testing. Feasibility indexes will be reported by descriptive statistics, such as mean with standard deviation and frequency with percentage. To test the hypothesis on the effects, a non-parametric test (i.e., Wilcoxon Signed-rank test) will be used to compare the outcome variables across time points to test the within-group effect in both groups separately. The level of significance was 0.05.

Significance: If this intervention is feasible and effective, this is going to provide a first of its kind home-based intervention to promote both cognitive functions and modify the dietary pattern of older people with cognitive frailty. First, it changes the cognitive training mode from a centre-based and supervised one to a home-based, self-paced, and tele-monitored one. Home-based training enables a more sustainable engagement of training for older people. This is particularly important during the COVID-19 pandemic period when all the elderly centres are closed. Home-based interventions are more accessible and convenient. It also solves the problem of space limitation in elderly centres in the community that more beneficiaries can be covered in space-limiting elderly centres. Second, it changes the mode of nutritional intervention from a supplement-based one to a daily-diet-based one. This intervention could enhance the nutrition and change their dietary pattern of community-dwelling older people with cognitive frailty by engaging them to protective diets, which ensures the sustainability of the beneficial effects of the protective diets towards cognitive frailty. Third, it changes the training mode from a training- and learning-oriented one to a gaming-oriented one. It brings more joy to community-dwelling older people even at the time when they are at home. It also fosters training adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years,
2. Community-dwelling, as defined by living at home without staying in long-term care facilities (e.g., nursing home) in the last 12 months as reported by the participants,
3. Cognitive frailty, as defined by co-existence of mild cognitive impairment and physical frailty,7

   1. Mild cognitive impairment, measured by Montreal Cognitive Assessment (MoCA) score ≤ 25 and Clinical Dementia Rating (CDR) score = 0.5,35,36 and
   2. Frailty status from pre-frail to frail, measured by Fried Frailty Phenotype score ≥ 1.37
4. Poor Mediterranean diet adherence, measured by MDS score < 30.5 (i.e., the mean MDS of community-dwelling older people reported in a local study),20 and
5. Functionally independent on food preparation, as defined by Lawton Instrumental Activity of Daily Living score ≥ 15/18 with the sub-score on Meal Preparation = 2/2.38,39

Exclusion Criteria:

1. Diagnosed dementia, according to subjects' medical record, or
2. Probable dementia, as defined by MoCA ≤ 18,35,36
3. Low vision (at least one eye with visual acuity < 20/60) or without corrective lens, because all training are visual-based and blurred vision negatively affects cognitive performance in cognitive training and assessment.40

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-05-14 (Estimated); Study Completion 2022-05-14 (Estimated)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet | Change is being assessed at 'baseline' (T0) and 'immediately after the completion of intervention' (T1), being 12 weeks apart
  Mediterranean diet was measured by the MedDietScore (MDS). The MDS covers two categories of items: beneficial foods (i.e., non-refined cereals, potatoes, fruits, vegetables, legumes, fish, and olive oil) and detrimental foods (i.e., red meat and products, poultry, full-fat dairy products, and alcohol). The MDS has demonstrated good criterion validity, showing a strong association with plasma and dietary fatty acids, and cardiovascular risks. Each MDS item is scored on a Likert scale from 0 to 5 to indicate the frequency of consumption, ranging from "never" to "daily" Summed MDS scores range from 0 to 55. A higher MDS indicates better adherence to the Mediterranean diet.

REFERENCES:
- [Derived] Kwan RYC, Law QPS, Tsang JTY, Lam SH, Wang KT, Sin OSK, Cheung DSK. The Effect of the Mediterranean Diet-Integrated Gamified Home-Based Cognitive-Nutritional (GAHOCON) Training Programme for Older People With Cognitive Frailty: Pilot Randomized Controlled Trial. JMIR Rehabil Assist Technol. 2024 Dec 13;11:e60155. doi: 10.2196/60155. PMID 39671585